CLINICAL TRIAL: NCT06871475
Title: The Effect Of Using Sticky Bone With Coronally Advanced Flap In Management Of Type 1 Gingival Recession
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ibrahim Abd Elhalim, researcher, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHDIRB2017122001
Record Dates: First submitted 2025-03-04; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): participant will receive sticky bone with coronally advanced flap
  Interventions: Biological: sticky bone with coronally advanced flap
- control group (Active Comparator): participants will undergo coronally advanced flap in treating gingival recession
  Interventions: Procedure: coronally advanced flap

INTERVENTIONS:
Biological: sticky bone with coronally advanced flap — using sticky bone with coronally advanced flap in treating the gingival recession
  Arms: study group
Procedure: coronally advanced flap — using coronally advanced flap alone in treating gingival recession
  Arms: control group

SUMMARY:
the main goal of this clinical trial is to evaluate the effect of sticky bone with coronally advanced flap in management of gingival recession in comparison to coronally advanced flap alone

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients of both sexes with age range 25-45 years old.
2. Patients are systemically healthy based on questionnaire dental modification of Cornell index.
3. O'Leary index (1972) is less than 10% (the surgical therapy is not initiated until the patient reaches the 10% level or less of plaque accumulation).
4. Buccal recession defects are classified RT1 according to Cairo's classification (2011).
5. Clinical indication and/or patient request for recession coverage.

Exclusion Criteria:

1. Pregnant female.
2. Smokers.
3. Patients with special needs or with any mental problems.
4. All patients are using any kind of medications that could interfere with healing of periodontal tissues. Such as chemotherapy and radiotherapy.
5. Teeth with carious lesions.
6. Rotated and extruded teeth.
7. Patient undergone any prior periodontal surgery in the relevant region within year.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
recession depth | changes in millimeters from base line up to 6 months
  is measured from CEJ to the gingival margin in millimeters.
thickness of keratinized gingiva | changes in biotype in millimeters from base line to follow up after 6 months
  thickness of the keratinized gingiva in the faciolingual direction (gingival biotype)

SECONDARY OUTCOMES:
Recession Width | changes in millimeters from base line to follow up after 6 months
  the widest point from the mesial gingival margin to the distal gingival margin in millimeters
the height of keratinized gingiva | changes in millimeters from base line up to 6 months
  the distance from the mucogingival junction to the gingival margin
percentage of root coverage | changes in percentile from base line up to 6 months
  it is the [pre-operative gingival recession depth - post-operative recession depth]/ [preoperative recession depth] * 100%
Probing pocket depth | changes in millimeters from base line up to 6 months
  the distance from the gingival margin to base of pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmonem Ebrahem, Professor, Study Chair — Minia University; Ahmed Abdallah Khalil, professor, Study Chair — Minia University; AyaAllah Kamal Abd El-al, lecturer, Study Director — Minia University; Shaimaa Mohamed Ibrahim, Principal Investigator — Minia University
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

REFERENCES:
- [Result] Ogata Y, Bui M, Griffin TJ, Hur Y. Use of Allograft with Platelet Concentrate in the Treatment of Multiple Miller Class III Gingival Recession Defects: Report of Three Cases. Int J Periodontics Restorative Dent. 2017 May/Jun;37(3):339-344. doi: 10.11607/prd.2673. PMID 28402343
- [Result] Wang HL, Kimble K, Eber R. Use of bone grafts for the enhancement of a GTR-based root coverage procedure: a pilot case study. Int J Periodontics Restorative Dent. 2002 Apr;22(2):119-27. PMID 12019707
- [Result] Sohn, D., B, H., J, K., Park WE, & Park CC. (2015). Utilization of autologous concentrated growth factors (CGF) enriched bone graft matrix(Sticky bone) and CGF-enriched fibrin membrane in implant dentistry. Jr Implant Adv Cli Dent.
- [Result] Mathur A, Jain M, Jain K, Samar M, Goutham B, Swamy PD, Kulkarni S. Gingival recession in school kids aged 10-15 years in Udaipur, India. J Indian Soc Periodontol. 2009 Jan;13(1):16-20. doi: 10.4103/0972-124X.51889. PMID 20376235
- [Result] Louis F. Rose, D. M. (2006). Surgical Therapies for the Treatment of Gingival Recession. Inside dentistry.
- [Result] Kimble KM, Eber RM, Soehren S, Shyr Y, Wang HL. Treatment of gingival recession using a collagen membrane with or without the use of demineralized freeze-dried bone allograft for space maintenance. J Periodontol. 2004 Feb;75(2):210-20. doi: 10.1902/jop.2004.75.2.210. PMID 15068108
- [Result] Hadziabdic, N. (2022). PRF and Sticky Bone as Regenerative Materials in Oral Surgery. IntechOpen. doi:10.5772/intechopen.108807
- [Result] Ghoderao D, Rathod S, Kolte AP, Bawankar P, Jadhav A. Randomized, controlled clinical trial to evaluate efficacy of sticky bone and concentrated growth factor in the management of intrabony defects: 12 months follow-up study. Dent Res J (Isfahan). 2022 Aug 16;19:67. eCollection 2022. PMID 36159047
- [Result] Kapa BP, N K S, G V G, Mehta DS. Coronally Advanced Flap Combined With Sticky Bone and i-PRF-Coated Collagen Membrane to Treat Single Maxillary Gingival Recessions: Case Series. Clin Adv Periodontics. 2022 Sep;12(3):147-151. doi: 10.1002/cap.10164. Epub 2021 May 15. PMID 33938633
- [Result] Chatterjee A, Sharma E, Gundanavar G, Subbaiah SK. Treatment of multiple gingival recessions with vista technique: A case series. J Indian Soc Periodontol. 2015 Mar-Apr;19(2):232-5. doi: 10.4103/0972-124X.145836. PMID 26015680